CLINICAL TRIAL: NCT05214781
Title: The Significance of Radiologically Detected Intramammary Lymph Nodes in Prediction of Axillary Lymph Nodes Status in Breast Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Collaborators: Mansoura University Hospital (Other)
Responsible Party: Principal Investigator, Ayman Shemes, Assistant lecturer of general surgery, Mansoura University
Other Study IDs: MD.21.09.521.R
Record Dates: First submitted 2022-01-04; First posted 2022-01-31 (Actual); Last update posted 2022-02-14 (Actual); Status verified 2022-01

CONDITIONS: Breast Neoplasms
Keywords: breast surgery , breast cancer , magnetic resonance image
MeSH Terms: conditions — Breast Neoplasms | interventions — Mastectomy, Modified Radical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: modified radical mastectomy — excision of the whole breast tissue including nipple and skin with axillary clearance
  Other Names: conservative breast surgey

SUMMARY:
Breast cancer is a major cause of mortality among women if not treated in early stages. Early screening and diagnosis have a lot to do with the therapeutic effect of prognosis .

Nodal status in breast cancer is one of the determining factors for staging, treatment, and prognosis. Nodal status in breast cancer is one of the determining factors for staging, treatment, and prognosis. Nodal status in breast cancer is one of the determining factors for staging, treatment, and prognosis .

Intramammary lymph nodes (IMLN) are defined as a lymph nodes that should be surrounded by breast tissue in all sides, which differentiate them from those in the axillary region .

Normal IMLN are typically described in all imaging study (mammography, ultrasound and magnetic resonance imaging [MRI]) as a circumscribed mass, smaller than 10 mm, with oval shape and hilar fat, usually at a peripheral location, adjacent to a vein . The most common location (about 70%) is the upper outer quadrants, however, it may be located anywhere in the breast .

DETAILED DESCRIPTION:
Aim of the work

* Primary outcome: prediction of axillary lymph nodes status by detection of Intramammary lymph nodes by radiological study.
* Secondary outcome: pathological correlation of molecular subtypes of breast cancer with radiological results.

Patients and Methods This is a prospective study, which will be conducted at Mansoura University Hospital from September 2021 till September 2023. This study will include thirty patients with breast cancer, after informed written consent taken from each case before being included in the study.

• Inclusion criteria included: Female patients aged more than 18 years old presented with breast cancer with radiologically detected intramammary lymph nodes and agreed to participate in the study.

• Exclusion criteria included:

1. Pregnancy.
2. Psychological instability.
3. Patients who refused to participate in our study.
4. Patients whose age less than 18 years old. * The enrolled patients will be subjected to:

1-preoperative assessment: Detailed history and clinical breast examination.

Investigations:

Laboratory :

Complete blood picture (CBC) Liver function test Kidney function test International normalized ratio (INR)

Radiology:

Bilateral breast ultrasonography. Digital mammography for patients > 40 years old. Breast Dynamic Contrast Enhanced and diffusion weighted magnetic resonance imaging.

5- Operative techniques: Modified radical mastectomy and conservative breast surgery with axillary clearance 6- Post-Operative follow up:

* Patient will stay in hospital for 1 to 2 days according to procedure and will be on antibiotic and analgesic according to hospital protocol.
* follow up amount and the color of fluid which discharge from drain.
* The wound is inspected after 48 h to be assessed.
* Histopathological examination of the specimen
* Immunohistochemistry will be done (estrogen receptor (ER) , progesterone receptor (PR) , HER-2neu and Ki-67 ) to determine the molecular subtypes of breast cancer
* We will correlate pathological data to radiological results.
* determine the post-operative type of systemic treatment according to pathological results.

ELIGIBILITY:
Inclusion Criteria:

* Female patients aged more than 18 years old presented with breast cancer with radiologically detected intramammary lymph nodes and agreed to participate in the study

Exclusion Criteria:

* Pregnancy.
* Psychological instability.
* Patients who refused to participate in our study.
* Patients whose age less than 18 years old.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a prospective study, which will be conducted at Mansoura University Hospital from September 2021 till September 2023. This study will include thirty patients with breast cancer, after informed written consent taken from each case before being included in the study.
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2021-09-14 (Actual); Primary Completion 2022-08-04 (Estimated); Study Completion 2023-03-04 (Estimated)

PRIMARY OUTCOMES:
prediction of axillary lymph nodes status | 6 months
  prediction of axillary lymph nodes status by detection of Intramammary lymph nodes by radiological study.

SECONDARY OUTCOMES:
pathological correlation | 7 months
  pathological correlation of molecular subtypes of breast cancer with radiological results.

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of medicine-Mansoura university - Egypt, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
This is a prospective study, which will be conducted at Mansoura University Hospital from September 2021 till September 2023. This study will include thirty patients with breast cancer, after informed written consent taken from each case before being included in the study.